CLINICAL TRIAL: NCT01929096
Title: Compound Edaravone Injection for Acute Ischemic Stroke, a Multi-center, Randomized, Double-blind, Multi-dose, Parallel, and Controlled Phase II Trial
Brief Title: Compound Edaravone Injection for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-23-01
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low-dose group (Experimental): Compound Edaravone Injection, 12.5mg/dose (Edaravone 10mg, (+)-Borneol 2.5mg), one dose every 12 hours, continue for 14 days
  Interventions: Drug: Compound Edaravone Injection
- Medium-dose group (Experimental): Compound Edaravone Injection, 37.5mg/dose (Edaravone 30mg, (+)-Borneol 7.5mg), one dose every 12 hours, continue for 14 days
  Interventions: Drug: Compound Edaravone Injection
- High-dose group (Experimental): Compound Edaravone Injection, 62.5mg/dose (Edaravone 50mg, (+)-Borneol 12.5mg), one dose every 12 hours, continue for 14 days
  Interventions: Drug: Compound Edaravone Injection
- Control group (Active Comparator): Edaravone Injection，30 mg/dose, one dose every 12 hours, continues for 14 days
  Interventions: Drug: Edaravone Injection

INTERVENTIONS:
Drug: Compound Edaravone Injection
  Arms: High-dose group; Low-dose group; Medium-dose group
Drug: Edaravone Injection
  Arms: Control group

SUMMARY:
1. To investigate the efficacy and safety of multi-doses Compound Edaravone Injection versus Edaravone Injection for acute ischemic stroke patients;
2. To provide evidence for the design of Compound Edaravone Injection Phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients, diagnosed of ischemic stroke;
* Onset of stroke is less than or equal to 48 hours;
* There are clear signs of neurological deficit: 4≤NIHSS score≤24, and also, the sum of NIHSS score for the upper limb and the lower limb is greater than or equal to 2;
* Patients signed written inform consent.

Exclusion Criteria:

* Cranial CT scan finds intracranial bleeding disorders: hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage;
* Iatrogenic stroke;
* Severe disturbance of consciousness: NIHSS category 1a for consciousness is greater than 1；
* The mRS score prior to this onset is greater than 1;
* Transient ischemic attack (TIA);
* SBP after blood pressure control is still greater than to equal to 220 mmHg, or DBP after blood pressure control is still greater than or equal to 120 mmHg;
* Patients with severe mental disorders and dementia;
* ALT or AST is greater than 2.0×ULN or previously known liver diseases, such as acute hepatitis, chronic active hepatitis, liver cirrhosis;
* Creatinine clearance is less than 30 ml/min or previously known severe renal diseases;
* Therapeutic neuroprotective agents have been applied after onset, including commercially available edaravone, nimodipine, ganglioside, citicoline, piracetam, butyl benzene peptides, Urinary Kallidinogenase;
* Arterial or venous thrombolytic therapy has been applied after onset;
* With malignant tumors or receiving concurrent antitumor treatment;
* With severe systemic disease, life expectancy is less than 90 days;
* Pregnant or lactating women;
* Participate in other clinical studies within 30 days before randomization;
* The investigators consider the patients are not suitable for this trial.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
mRS score on day 90 | day 90
Change from baseline NIHSS score on day 14 | day 14

SECONDARY OUTCOMES:
The proportion of patients with NIHSS score 0-1 (including motor function) on day 14, 30, 90 | day 14, 30, 90
The proportion of patients with Barthel Index (BI) score greater than or equal to 95 on day 14, 30, 90 | day 14, 30, 90
The Montreal Cognitive Assessment(MoCA) score on day 14, 30, 90 | day 14, 30, 90
Stroke Impact Scale (SIS) score on day 90 | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (28):
- China (28):
  - Navy General Hospital of The Chinese PLA, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Third Military Medical University of Chinese PLA, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Haerbin Medical University, Haerbin, Heilongjiang
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Central Hospital of Baotou, Baotou, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The General Hospital of Shenyang Military, Chinese PLA, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Xu J, Wang Y, Wang A, Gao Z, Gao X, Chen H, Zhou J, Zhao X, Wang Y. Safety and efficacy of Edaravone Dexborneol versus edaravone for patients with acute ischaemic stroke: a phase II, multicentre, randomised, double-blind, multiple-dose, active-controlled clinical trial. Stroke Vasc Neurol. 2019 Apr 22;4(3):109-114. doi: 10.1136/svn-2018-000221. eCollection 2019 Sep. PMID 31709115